CLINICAL TRIAL: NCT02781207
Title: Comparison Between Standard and Bedside Ultrasound Integrated Approach for Risk Stratification of Patients Presenting With Syncope in the Emergency Department
Brief Title: Comparison Between Standard and Ultrasound Integrated Approach for Risk Stratification of Syncope in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Enrico Lupia, MD, PhD, Associate Professor, MD, PhD, University of Turin, Italy
Other Study IDs: unito_isyncope
Record Dates: First submitted 2016-05-11; First posted 2016-05-24 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Syncope
Keywords: syncope; point-of-care ultrasound
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a observational prospective study. For patients presenting to the Emergency Department with loss of consciousness, emergency physicians will be asked to screen the real syncope without an evident and immediate cause for the loss of consciousness (e.g. vasovagal) and/or at least one high risk condition as listed by the European Society of Cardiology in the 2009 Guidelines for the diagnosis and management of syncope (i.e. severe structural or coronary artery disease, clinical or ECG features suggesting arrhythmic syncope, and important co-morbidities).

In case of a real syncope not clearly physiopathologically explained and no high risk conditions, the emergency physician in charge will check risk factors for high risk syncope and categorize again every cases.

A high risk syncope is characterized by at least one high-risk characteristic (based on 2015 "Syncope clinical management in the emergency department consensus"): syncope during exertion, in supine position, with new onset of chest discomfort, palpitations before the loss of consciousness, family history of sudden death, congestive heart failure, aortic stenosis, left ventricular outflow tract disease, dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, left ventricular ejection fraction <35%, previously documented ventricular arrhythmia, coronary artery disease, congenital heart disease, previous myocardial infarction, pulmonary hypertension, previous ICD implantation, anemia (i.e. Hb <9 g/dl), lowest systolic blood pressure in the ED <90 mmHg, sinus bradycardia (<40 bpm), new (or previously unknown) left bundle branch block, bifascicular block plus a first degree AV block, Brugada ECG pattern, ECG changes consistent with acute ischemia, a new non-sinus rhythm, bifascicular block, and a prolonged QTc (>450 ms).

Low and intermediate risk syncopes will be enrolled and evaluated using an integrated point-of-care sonographic approach (based on history, physical exam, electrocardiogram, and lung, focus cardiac and venous compression ultrasonography).

After discharge, the risk of patient's syncope will be determined by reviewing the entire medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients evaluated in the Emergency Department for loss of consciousness

Exclusion Criteria:

* identification of cause of loss of consciousness after initial evaluation;
* loss of consciousness classified as high risk syncope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort is composed of all adult patients evaluate in the Emergency Department for syncope (defined as transient loss of consciousness due to global cerebral hypoperfusion characterized by rapid onset, short duration, and spontaneous complete recovery, and unrelated to trauma).
  After first evaluation, high risk syncope will be excluded.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
number of low risk acute syncope reclassified to intermediate/high risk after integrated point-of-care ultrasound evaluation | during the stay in the Emergency Department (ideally within 6 hours or, if patient will be admitted in the observational unit ward, within 36 hours)
number of intermediate risk acute syncope reclassified to low risk after integrated point-of-care ultrasound evaluation | during the stay in the Emergency Department (ideally within 6 hours or, if patient will be admitted in the observational unit ward, within 36 hours)
number of intermediate risk acute syncope reclassified to high risk after integrated point-of-care ultrasound evaluation | during the stay in the Emergency Department (ideally within 6 hours or, if patient will be admitted in the observational unit ward, within 36 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: Yes
The study collect only clinical data, also reported in the Emergency Department chart. The chart is always given to the patient at the discharge.